CLINICAL TRIAL: NCT00124722
Title: A Randomized, Assessor-blind, Dose-ranging, Phase IIIB, Multicenter Trial Comparing the Intubating Conditions and Time Course of Block of Three Different Intubating Doses (0.45 mg/kg, 0.6 mg/kg, and 1.0 mg/kg) of Zemuron® in Pediatric and Adolescent Subjects Under General Anesthesia
Brief Title: A Study to Compare Different Intubating Doses of Zemuron in Pediatric and Adolescent Subjects Under General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05798; 021049
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.45 mg/kg Zemuron (Experimental): 0.45 mg/kg Zemuron
  Interventions: Drug: Rocuronium bromide (Zemuron)
- 0.6 mg/kg Zemuron (Active Comparator): 0.6 mg/kg Zemuron
  Interventions: Drug: Rocuronium bromide (Zemuron)
- 1.0 mg/kg Zemuron (Experimental): 1.0 mg/kg Zemuron
  Interventions: Drug: Rocuronium bromide (Zemuron)

INTERVENTIONS:
Drug: Rocuronium bromide (Zemuron) — A single IV Zemuron bolus dose of 0.45 mg/kg prior to intubation.
  Other Names: ORG 9426; SCH 900085; Zemuron
  Arms: 0.45 mg/kg Zemuron
Drug: Rocuronium bromide (Zemuron) — A single IV Zemuron bolus dose of 0.6 mg/kg prior to intubation.
  Other Names: ORG 9426; SCH 900085; Zemuron
  Arms: 0.6 mg/kg Zemuron
Drug: Rocuronium bromide (Zemuron) — A single IV Zemuron bolus dose of 1.0 mg/kg prior to intubation.
  Other Names: ORG 9426, SCH 900085, Zemuron
  Arms: 1.0 mg/kg Zemuron

SUMMARY:
The primary purpose of this study is to evaluate the time course of muscle relaxation after administration of three different single intravenous bolus doses of rocuronium bromide for intubation (insertion of a tube through the nose or mouth into the trachea to provide artificial ventilation) in term neonates (birth to <28 days old), infants (28 days to <=3 months) and toddlers (>3 months to <=2 years), children (2 years to less than or equal to 11 years of age), and adolescents (>11 years to less than or equal to 17 years of age).

Subjects in each of the age groups will be randomized to one of 3 Zemuron® doses: 0.45 mg/kg, 0.6 mg/kg, or 1.0 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects from birth up to 17 years of age who will be scheduled for surgery under general anesthesia.

Exclusion Criteria:

* Subjects whose parent(s) or legal guardian(s) are not willing to give written consent and where applicable, subjects who have not given appropriate assent to participate in the trial will not be allowed to enter.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time to reappearance of T3 (time from end-administration of Zemuron to reappearance of the third twitch of a TOF stimulation) | during surgery

SECONDARY OUTCOMES:
Onset time, maximum block, time to reappearance of T1, Recovery to TOF 0.7, 0.8 and 0.9 and intubation score | during and after surgery

REFERENCES:
- [Result] Tirotta CF, Brandom B, Siddiqui MS, Ehlers M, Betzel J, Chen J-Y, De Bie J, Blobner M. Time Course of Rocuronium-Induced Neuromuscular Blockade in Pediatric Patients: A Phase III, Randomized, Dose-Response Study. J Anesthe Clin Res. 2012;3:189.